CLINICAL TRIAL: NCT06803680
Title: A Phase 1, Open-Label Study Investigating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Antitumor Activity of BGB-B455 in Patients With Selected Advanced or Metastatic Solid Tumors
Brief Title: A Study of BGB-B455 in Adults With Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BGB-B455-101; 2024-512931-64-00 (EU CTIS Number); CTR20251939 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor
Keywords: Claudin-6; CLDN6+; advanced or metastatic solid tumor; CD3; BsAb; bispecific antibody; CD3-BsAb; CLDN
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1a: Dose Escalation and Safety Expansion (Experimental): Sequential cohorts of increasing dose levels of BGB-B455 will be evaluated as monotherapy.
  Interventions: Drug: BGB-B455
- Phase 1b: Dose Expansion (Experimental): Recommended Dose(s) for Expansion (RDFE[s]) of BGB-B455 determined from Phase 1a as monotherapy or in combination with investigator-selected chemotherapy will be evaluated for selected indications based on emerging data.
  Interventions: Drug: BGB-B455; Drug: Chemotherapy

INTERVENTIONS:
Drug: BGB-B455 — Planned doses administered on specified days per protocol.
Drug: Chemotherapy — Administered in accordance with relevant local guidelines and/or prescribing information.
  Arms: Phase 1b: Dose Expansion

SUMMARY:
The goal of this clinical trial is to learn if BGB-B455 can treat advanced or metastatic solid tumors expressing claudin 6 (CLDN6), a protein that is found on some tumors.

The main questions it aims to answer are:

* What is the recommended dosing for BGB-B455?
* What medical problems do participants have when taking BGB-B455?

The study has two parts:

* Phase 1a: dose escalation and safety expansion
* Phase 1b: dose expansion

DETAILED DESCRIPTION:
Claudin proteins are cell proteins that can play an important role in how cancer starts and progresses. Because of its preferential expression in tumors compared to normal tissues, CLDN6 is an ideal tumor antigen to target for treatment. BGB-B455 is a bispecific antibody (BsAbs) that targets CLDN6 on tumor cells and the CD3 receptor on T cells, which may provide a CLDN6-dependent antitumor immune response in a more tolerable manner without undue systemic toxicity.

This new study will check how safe and helpful this potential anticancer drug is. In addition, this study will explore the recommended dosing level for BGB-B455. This drug will be tested by itself or in combination with investigator-selected chemotherapy in participants with selected solid tumors expressing the CLDN6 protein.

This study is an open label study, meaning that both you and your study doctor will know what study drug/treatment you are given. This study has two parts:

* Phase 1a consists of a dose escalation part where increasing amounts of the study treatment are given to different dose cohorts, and a safety expansion part that will enroll additional participants at selected doses for further assessments.
* Phase 1b (dose expansion) will enroll participants at the best dose found in Phase 1a to see if it helps people with certain solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced or metastatic, and unresectable solid tumors who have previously received standard systemic therapy for advanced or metastatic disease or for whom treatment is not available or not tolerated.
* Agreement for collection of formalin-fixed paraffin-embedded (FFPE) tumor tissue for central CLDN6 testing and other biomarker assessments.
* Tumor CLDN6 expression (CDLN6+) by central immunohistochemistry testing is required for certain cohorts.
* ≥ 1 measurable lesion as assessed by RECIST v1.1.
* Stable Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Adequate organ function.

Exclusion Criteria:

* Prior systemic anticancer therapy, including chemotherapy, immunotherapy (eg, interleukin, interferon, thymosin), targeted therapy, and antibody drug conjugates (ADCs) that are standard or investigational agents (including herbal medicine or Chinese [or other country] patent medicines, ≤ 14 days or 5 half-lives (whichever is shorter) before the first dose of study drug(s).
* Palliative radiation treatment or other locoregional therapies ≤ 14 days before the first dose of study drug(s).
* Live vaccine ≤ 28 days before the first dose of study drug(s). Vaccines for COVID-19 are allowed except for any live vaccine that may become available. Seasonal vaccines for influenza are generally inactivated vaccines and are allowed. Intranasal vaccines are live vaccines and are not allowed.
* Any major surgical procedure ≤ 28 days before the first dose of study drug(s).
* History of prior ≥ Grade 3 cytokine release syndrome (CRS).
* Participants with toxicities (because of prior anticancer therapy) that have not recovered to baseline or stabilized, except for adverse events not considered a likely safety risk (eg, alopecia, neuropathy, and specific laboratory abnormalities).

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Number of participants with adverse events (AEs) and serious adverse events (SAEs) | From the first dose of study drug(s) to 30 days after the last dose or initiation of a new anticancer therapy, whichever occurs first; up to approximately 7 months
  Number of participants with AEs and SAEs, including laboratory abnormalities, and AEs that meet protocol-defined dose-limiting toxicity (DLT) criteria or protocol-defined adverse events of special interest (AESI) criteria.
Phase 1a: Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD) of BGB-B455 | Approximately 1 month
  MTD is defined as the highest dose evaluated for which estimated toxicity rate is the closest to the target toxicity rate. MAD is defined as the highest dose administered if MTD is not reached.
Phase 1a: RDFE of BGB-B455 | Approximately 1 month
  RDFE of BGB-B455 will be determined based upon the MTD or MAD.
Phase 1b: Overall Response Rate (ORR) | Approximately 18 months
  ORR is defined as the percentage of participants with best overall response of complete response (CR) or partial response (PR), as determined from tumor assessments by investigator per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). CR and PR must be confirmed by repeat assessments.

SECONDARY OUTCOMES:
Phase 1a: ORR | Approximately 18 months
  ORR is defined as the percentage of participants with best overall response of CR or PR, as determined from tumor assessments by investigator per RECIST v1.1. CR and PR must be confirmed by repeat assessments.
Phase 1a and 1b: Duration of Response (DOR) | Approximately 18 months
  DOR is defined as the time from the first confirmed objective response to documented disease progression or death, whichever occurs first, as determined from tumor assessments by investigator per RECIST v1.1.
Phase 1a and 1b: Disease Control Rate (DCR) | Approximately 18 months
  DCR is defined as the percentage of participants who achieve CR, PR, or stable disease, as determined from tumor assessments by investigator per RECIST v1.1.
Phase 1a and 1b: Time to Response (TTR) | Approximately 18 months
  TTR is defined as the time from the date of the first administration of study drug to the first confirmed response, as determined from tumor assessments by investigator per RECIST v1.1.
Phase 1a and 1b: Serum concentrations of BGB-B455 | Approximately 7 months
Phase 1a and 1b: Number of participants with anti-drug antibodies (ADAs) to BGB-B455 | Approximately 7 months
Phase 1b: Progression-Free Survival (PFS) | Approximately 18 months
  PFS is defined as the time from the date of the first administration of study drug to the date of the first documentation of disease progression or death, whichever occurs first, as determined from tumor assessments by investigator per RECIST v1.1.
Phase 1b: Number of participants with AEs | From the first dose of study drug(s) to 30 days after the last dose or initiation of a new anticancer therapy, whichever occurs first; up to approximately 7 months
  Number of participants with AEs, including physical examinations, electrocardiograms (ECGs), and laboratory assessments as indicated.
Phase 1a and 1b: Area under the concentration-time curve (AUC) of BGB-B455 | Approximately 4 months
Phase 1a and 1b: Maximum observed plasma concentration (Cmax) of BGB-B455 | Approximately 4 months
Phase 1a and 1b: Time to reach maximum observed plasma concentration (Tmax) of BGB-B455 | Approximately 4 months
Phase 1a and 1b: Trough Concentration (Ctrough) of BGB-B455 | Approximately 7 months
Phase 1a and 1b: Apparent clearance (CL) of BGB-B455 | Approximately 4 months
Phase 1a and 1b: Volume of distribution (Vd) of BGB-B455 | Approximately 4 months
Phase 1a and 1b: Accumulation Ratio of BGB-B455 | Approximately 4 months
Phase 1a and 1b: Terminal half-life (t1/2) of BGB-B455 | Approximately 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (14):
- United States (6):
  - Adventhealth, Celebration, Florida
  - Florida Cancer Specialists and Research Institute, Lake Mary, Florida
  - Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Next Oncology, Austin, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Australia (3):
  - Blacktown Cancer and Haematology Centre, Blacktown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Mater Cancer Care Centre, South Brisbane, Queensland
- China (5):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Sun Yat Sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - Fudan University Shanghai Cancer Centerpudong, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/